CLINICAL TRIAL: NCT00067600
Title: Lifestyle Changes to Increase Bone Density in Teen Girls
Brief Title: Improving Bone Health in Adolescent Girls: The Youth Osteoporosis and Understanding Total Health (YOUTH) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: R01HD037744 (NIH)
Record Dates: First submitted 2003-08-25; First posted 2003-08-26 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Diet; Vegetables; Calcium; Resistance Training

INTERVENTIONS:
Behavioral: Diet with increased fruits, vegetables, and calcium
Behavioral: Increased high impact activity and resistance training

SUMMARY:
Osteoporosis affects nearly half of all American women over age 50. During the teenage years, girls can increase bone growth to decrease their risk of osteoporosis later in life. This study will test whether girls can change their food intake and physical activity patterns in ways that will increase their bone growth during the mid-teen years.

DETAILED DESCRIPTION:
Osteoporosis-related fractures incur an annual cost in the United States of more than $8 billion. Peak bone mass is achieved in the late teens and early 20s. An important component of a lifelong osteoporosis prevention strategy is to maximize bone mineral content during the teen years and establish lifestyle patterns that will help maintain bone mineral content through menopause. This trial will test the efficacy of a comprehensive lifestyle intervention to build bone and prevent bone loss among adolescent women 14 to 16 years of age.

Participants in this study will be randomized to either an intervention group or an attention control group. The intervention program includes a physical activity component involving high impact and spinal motion activities and a diet component rich in fruits, vegetables, and calcium. Participants will take part in group and individual meetings and activities and receive coaching telephone calls. Participants will be assessed at study entry and two annual follow-up visits. Primary outcome measures include objective measures (serum folate and carotenoids urinary sodium, lean body mass, accelerometer measure of physical activity) and self-reports.

ELIGIBILITY:
Inclusion Criteria

* High school freshman or sophomore
* Body mass index (BMI) from 16 through 23
* Member of Kaiser Permanente Northwest Health Plan
* Parent or guardian willing to participate

Exclusion Criteria

* Co-morbidity requiring a specific diet
* Medication which contraindicates consuming a high-fiber diet
* Life-threatening disease or other condition that would interfere with study participation
* Current or past medically or self-diagnosed eating disorder
* Current behaviors consistent with eating-related disorder
* Pregnancy
* Diagnosis of psychological disorder or difficulty within the past year

Ages: 14 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 228
Dates: Start 2000-08; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Total Body Bone Mineral Density (TBBMD) | Baseline, 1 year, and 2 years
  Changes in TBBMD as measured by DEXA at baseline, 1 year, and 2 years

SECONDARY OUTCOMES:
Serum osteocalcin, alkaline phosphatase, and urinary n-telopeptide | Baseline, 1 year, and 2 years
  Biologic measures of bone metabolism
Plasma carotenoids and red cell folate | Baseline, 1 year, and 2 years
  Biologic measures of dietary change

CONTACTS AND LOCATIONS:
Overall Officials: Lynn L DeBar, PhD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States

REFERENCES:
- [Derived] DeBar LL, Ritenbaugh C, Aickin M, Orwoll E, Elliot D, Dickerson J, Vuckovic N, Stevens VJ, Moe E, Irving LM. Youth: a health plan-based lifestyle intervention increases bone mineral density in adolescent girls. Arch Pediatr Adolesc Med. 2006 Dec;160(12):1269-76. doi: 10.1001/archpedi.160.12.1269. PMID 17146025